CLINICAL TRIAL: NCT01671917
Title: Evaluation of an Educational Program Associated With Exercises (EDEX) Before Total Knee Arthroplasty
Acronym: EDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Paris 5 - Rene Descartes (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOM 10042
Record Dates: First submitted 2012-07-20; First posted 2012-08-24 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Total knee replacement; Knee osteoarthritis; Education; Exercise; Handicap; Function; Cost-effectiveness; Cost-utility; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational and exercise program (Experimental)
  Interventions: Other: Educational and exercise program
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Educational and exercise program — * 4 (twice a week) group education sessions lasting 30 minutes plus an education booklet about knee replacement
  * 4 (twice a week) sessions of an exercise programme lasting 1 hour
  Arms: Educational and exercise program
Other: Usual care — Information and counseling usually provided in orthopedics department and an information booklet about knee replacement.
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether a standardized education and exercise program proposed before a total knee replacement for knee osteoarthritis is effective in functional recovery after surgery.

DETAILED DESCRIPTION:
Knee osteoarthritis leads to deficiencies in muscle strength, knee range of motion and balance, and cardio respiratory deconditioning that contribute to alter abilities to perform activities of daily living. It is the principal indication for total knee arthroplasty (TKA). Patients' functional state and pain level are generally improved after TKA and the physical and functional status pre-TKA are predictive of recovery after surgery. Decreasing length of stay at surgery departments and promoting return at home after TKA are recommended. The recommendations of the Health Authority in France (HAS) and the new law of finance for French clinics contribute to shorter hospital stays and to restrain the conditions of admission to Physical Medicine and Rehabilitation department after TKA.Exercise and education programs conducted before TKA could help better prepare patients for surgery, improve functional outcome and accelerate functional recovery after surgery thus reducing the length of stay in orthopedic departments and facilitate return to home (directly or after a stay in PMR departments). The type of program necessary to achieve those goals remains to be defined.A systematic review of the literature associated with an analysis of practices about the relevance of rehabilitation programs before TKA, concluded that the implementation of such programs before TKA was likely to reduce the length of stay in surgery departments and improve the rate of direct return to home after surgery but that high quality trials were lacking. It also suggested that association of exercise programs with educational ones could be more effective than exercise or education alone, particularly for fragile patients with impaired functional capacity, co-morbidities and/or social problems.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 50 to 85 years
* Patient suffering from knee osteoarthritis according to ACR for which a total knee arthroplasty is scheduled
* Preliminary medical examination whose results will be transmitted to the patient
* Patient giving his informed consent to participate in the study
* Patient affiliated to or beneficiary of social insurance

Exclusion Criteria:

* Patients institutionalized
* Patients who have already received an ipsilateral total knee arthroplasty
* Patients with chronic inflammatory arthritis
* Cognitive or behavioral disorders making assessment impossible
* Inability to speak and write French
* TKA indicated for other reason than osteoarthritis

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
The percentage of patients able to quit independently the orthopedic department | at day 4 post-surgery
  Assessed by the ability to perform lying-sitting and sitting-standing transfers, walk 30 meters and go up and down one floor at day 4 (± 1 day) after the surgery. Each item will be scored on a 4-class scale (0, unable to perform and 3, able to perform independently). Ability to quite the orthopedic department will be defined as scoring 3 out of 3 for all 4 assessed items on the day of discharge from the orthopedic department.
Changes from baseline in functional recovery | 6 months post-surgery
  Assessed by the area under the curve of the function subscale of the WOMAC index within the first 6 months post-surgery

SECONDARY OUTCOMES:
Changes from baseline in mean knee pain in the previous 48 hrs | 6 months post-surgery
  Assessed by a self-administered 11-point numeric rating scale (0, no pain and 100, maximal pain)
Changes from baseline in mean knee pain in the previous 48 hrs | 12 months post-surgery
  Assessed by a self-administered 11-point numeric rating scale (0, no pain and 100, maximal pain)
Changes from baseline in mean function in the previous 48 hrs | 6 months post-surgery
  Assessed by the self-administered WOMAC function subscale (0, best function and 100, worse function)
Changes from baseline in mean function in the previous 48 hrs | 12 months post-surgery
  Assessed by the self-administered WOMAC function subscale (0, best function and 100, worse function)
Changes from baseline in mean quality of life | 6 months post-surgery
  Assessed by the physical and mental components of the self-administered SF-12 questionnaire (0, worse quality of life and 100, best quality of life) and by the self-administered EQ-5D-3L questionnaire (11111, best quality of life and 33333, worse quality of life)
Changes from baseline in mean quality of life | 12 months post-surgery
  Assessed by the physical and mental components of the self-administered SF-12 questionnaire (0, worse quality of life and 100, best quality of life) and by the self-administered EQ-5D-3L questionnaire (11111, best quality of life and 33333, worse quality of life)
Changes from baseline in the mean number of steps in the previous week | 6 months post-surgery
  Assessed by the self-reported number of steps monitored by a podometer
Changes from baseline in the mean number of steps in the previous week | 12 months post-surgery
  Assessed by the self-reported number of steps monitored by a podometer
Satisfaction with the treatment | 6 months post-surgery
  Assessed by a self-administered 11-point numeric rating scale (0, not satisfied and 100, totally satisfied)
Satisfaction with the treatment | 12 months months post-surgery
  Assessed by a self-administered 11-point numeric rating scale (0, not satisfied and 100, totally satisfied)
Cost-effectiveness | 6 months post-surgery
  Assessed by the cost-utility ratio
Cost-effectiveness | 12 months months post-surgery
  Assessed by the cost-utility ratio
Adverse events | 12 months post-surgery
  Assessed by self reporting using an open-ended question

CONTACTS AND LOCATIONS:
Overall Officials: François Rannou, MD, PhD, Principal Investigator — AP-HP, Descartes University, INSERM; Pascal Richette, MD, PhD, Principal Investigator — CHU Lariboisière; Emmanuel Coudeyre, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Cochin, Paris, France

REFERENCES:
- [Background] Nguyen C, Boutron I, Roren A, Anract P, Beaudreuil J, Biau D, Boisgard S, Daste C, Durand-Zaleski I, Eschalier B, Gil C, Lefevre-Colau MM, Nizard R, Perrodeau E, Rabetrano H, Richette P, Sanchez K, Zalc J, Coudeyre E, Rannou F. Effect of Prehabilitation Before Total Knee Replacement for Knee Osteoarthritis on Functional Outcomes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e221462. doi: 10.1001/jamanetworkopen.2022.1462. PMID 35262716